CLINICAL TRIAL: NCT00770120
Title: Phase II Trial of mTOR Inhibitor, Everolimus (RAD001), in Malignant Pleural Mesothelioma (MPM)
Brief Title: S0722: Everolimus in Treating Patients With Pleural Malignant Mesothelioma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000616162; S0722 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Malignant Mesothelioma
Keywords: recurrent malignant mesothelioma; stage II malignant mesothelioma; stage III malignant mesothelioma; stage IV malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): Daily oral Everolimus 10 mg/day
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well everolimus works in treating patients with pleural malignant mesothelioma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the 4-month progression-free survival in patients with unresectable malignant pleural mesothelioma treated with everolimus.

Secondary

* To determine the response rate (confirmed and unconfirmed, complete and partial responses) and disease control rate (response or stable disease) in patients with measurable disease by RECIST and modified RECIST criteria.
* To determine overall survival of these patients.
* To evaluate the frequency and severity of toxicities associated with this treatment regimen.

OUTLINE: This is a multicenter study.

Patients receive oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant pleural mesothelioma

  * Unresectable disease
* Must have measurable or nonmeasurable disease by RECIST or modified RECIST criteria
* Must have received prior systemically administered* platinum-based chemotherapy and meets the following criteria:

  * No more than 2 prior systemic therapeutic regimens allowed (including biologics, targeted, and immunotherapies)
  * At least 1 regimen must have been platinum-based
  * Neoadjuvant and/or adjuvant systemic therapy is not counted as a prior regimen, assuming ≥ 12 weeks have elapsed between the end of neoadjuvant/adjuvant therapy and development of progressive disease NOTE: *Pleural space washing with cisplatin does not constitute systemic administration
* No known CNS metastases

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Serum bilirubin normal
* AST or ALT ≤ 1.5 times upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No evidence of bleeding diathesis or coagulopathy

  * Previous pulmonary embolism allowed provided the patient is on therapeutic low molecular weight heparin injections or warfarin AND no evidence of bleeding

    * Patients on therapeutic warfarin must have an INR of < 5 within 28 days prior to registration
* No pathologic condition other than mesothelioma that carries a high risk of bleeding
* No known HIV positivity
* No gastrointestinal tract disease resulting in an inability to take oral or enteral medication via a feeding tube or a requirement for IV alimentation, or active peptic ulcer disease
* No other prior malignancy allowed except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer from which the patient is currently in complete remission
  * Any other cancer from which patient has been disease-free for 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* At least 28 days since prior systemic therapy (42 days for nitrosoureas or mitomycin C)
* At least 28 days since prior thoracic or other major surgery (e.g., pleurectomy or pleurodesis) and no anticipated need for major surgical procedures during study
* At least 14 days since prior radiotherapy
* No prior surgical procedure affecting absorption
* No prior chronic, systemic corticosteroids or other immunosuppressive agent, except corticosteroids equivalent to prednisone ≤ 20 mg daily

  * Must have been on a stable dosage regimen for ≥ 4 weeks
  * Topical and inhaled corticosteroids allowed
* No prior mTOR inhibitor therapy (i.e., rapamycin, everolimus, or temsirolimus)
* No concurrent immunization with attenuated live vaccines
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent investigational therapy
* No other concurrent anticancer agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sai-Hong I. Ou, MD, PhD, Study Chair — Chao Family Comprehensive Cancer Center; Linda Garland, MD, Study Chair — University of Arizona
Locations (129):
- United States (129):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - University of California Davis Cancer Center, Sacramento, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - U.T. Medical Center Cancer Institute, Knoxville, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Ou SH, Moon J, Garland LL, Mack PC, Testa JR, Tsao AS, Wozniak AJ, Gandara DR. SWOG S0722: phase II study of mTOR inhibitor everolimus (RAD001) in advanced malignant pleural mesothelioma (MPM). J Thorac Oncol. 2015 Feb;10(2):387-91. doi: 10.1097/JTO.0000000000000360. PMID 25611229

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus: Daily oral Everolimus 10 mg/day
  everolimus
Period: Overall Study
Arm/Group | Everolimus
Started | 61
Eligible | 60
Not Analyzable | 1
Completed | 0
Not Completed | 61
Not completed — Progression | 31
Not completed — Adverse Event | 11
Not completed — Not Protocol Specified | 11
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Ineligible | 1
Not completed — Never Received Treatment/Not Analyzable | 1
Not completed — Reason under Review | 1

BASELINE CHARACTERISTICS:
Population: Number of patients who were eligible and received treatment and thus analyzable.
Arm/Group | Everolimus
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 67 [45.8 to 81.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 55
  More than one race | 0
  Unknown or Not Reported | 3
Histology [Number; unit: participants]
  Epithelial | 36
  Mesothelioma, NOS | 17
  Biphasic | 4
  Not Reported | 2
Number of Metastatic Sites [Number; unit: participants]
  None | 5
  Single | 23
  Multiple | 31
Prior Systemic Regimens [Number; unit: participants]
  1 Regimen | 34
  2 Regimens | 25
Performance Status [Number; unit: participants] — 0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  participants
    0 | 13
    1 | 46
Weight Loss Last 6 Months [Number; unit: participants]
  < 5% | 47
  5% - < 10% | 6
  10% - 20% | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-Free Survival was defined as the duration from the date of registration until the date of disease progression per RECIST or death due to any cause. Patients known to be alive without evidence of disease progression were censored at the date of last contact. Disease progression was defined as a >= 20% increase over nadir in the sum of longest diameters of target lesions, unequivocal progression of non-target lesions in the opinion of the treating investigator, appearance of new lesions, symptomatic deterioration, or death due to disease
Time Frame: Every 8 weeks until disease progression, up to 3 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 59
months | 3.0 [1.8 to 3.6]

2. Secondary Outcome: Response
Description: A response was defined as either a confirmed or unconfirmed complete or partial responses as defined by RECIST. A complete response (CR) was defined as the disappearance of all disease. A partial response (PR) was defined as a >= 30% decrease in the sum of longest diameters of target lesions. A CR or PR was considered confirmed if two consecutive determinations were made at least 4 weeks apart.
Time Frame: Every 8 weeks until disease progression, up to 3 years.
Measure: Number (95% Confidence Interval); unit: percentage of overall response rate
Arm/Group | Everolimus
Number analyzed (Participants) | 45
percentage of overall response rate | 2 [0 to 12]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the duration between the date of enrollment and the date of death due to any cause. Patients last known to be alive were censored at the date of last contact.
Time Frame: Every 8 weeks until disease progression, up to 3 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 59
months | 6.3 [4.8 to 8]

4. Secondary Outcome: Frequency and Severity of Toxicities
Time Frame: Weekly during the first 8 weeks of treatment, then every 4 weeks while on treatment, then every 8 weeks until disease progression, then every 6 months thereafter.
Population: Number of Subjects With Greater Than Grade 2 Toxicity
Measure: Number; unit: participants
Arm/Group | Everolimus
Number analyzed (Participants) | 59
participants
  Anorexia | 1
  Confusion | 1
  Dehydration | 2
  Diarrhea | 1
  Dyspnea (shortness of breath) | 3
  Fatigue (asthenia, lethargy, malaise) | 6
  Glucose, serum-high (hyperglycemia) | 3
  Hemoglobin | 4
  INR (of prothrombin time) | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 1
  Infection with unknown ANC - Lung (pneumonia) | 3
  Left ventricular systolic dysfunction | 1
  Lymphopenia | 2
  Mucositis/stomatitis (clinical exam) - Oral cavity | 1
  Mucositis/stomatitis (functional/symp) - Oral cav | 1
  Muscle weakness, not d/t neuropathy - body/general | 2
  Pneumonitis/pulmonary infiltrates | 2
  Rash/desquamation | 1
  Triglyceride, serum-high (hypertriglyceridemia) | 2

ADVERSE EVENTS:
Time Frame: From date of registration to 3 years post registration or death (whichever occurs first).
Description: All SAEs and AEs.
Arm/Group | Everolimus
Serious Adverse Events (participants affected / at risk) | 25/59
Other Adverse Events (participants affected / at risk) | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=59)
Hemoglobin (Blood and lymphatic system disorders) | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 5
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 4
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Confusion (Psychiatric disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 4
Thrombosis/thrombus/embolism (Vascular disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=59)
Hemoglobin (Blood and lymphatic system disorders) | 38
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 4
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 14
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Gastrointestinal-Other (Gastrointestinal disorders) | 5
Hemorrhoids (Gastrointestinal disorders) | 3
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 19
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 21
Pain - Abdomen NOS (Gastrointestinal disorders) | 9
Pain - Oral cavity (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 10
Constitutional Symptoms-Other (General disorders) | 3
Edema: limb (General disorders) | 8
Edema: trunk/genital (General disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 41
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 4
Pain - Chest/thorax NOS (General disorders) | 8
Pain-Other (General disorders) | 4
Rigors/chills (General disorders) | 4
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 5
AST, SGOT (Investigations) | 8
Alkaline phosphatase (Investigations) | 6
Cholesterol, serum-high (hypercholesterolemia) (Investigations) | 19
Creatinine (Investigations) | 14
Leukocytes (total WBC) (Investigations) | 12
Lymphopenia (Investigations) | 9
Metabolic/Laboratory-Other (Investigations) | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4
Platelets (Investigations) | 16
Weight loss (Investigations) | 16
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 15
Anorexia (Metabolism and nutrition disorders) | 27
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 6
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 26
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 30
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 7
Pain - Back (Musculoskeletal and connective tissue disorders) | 5
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 6
Neuropathy: sensory (Nervous system disorders) | 10
Pain - Head/headache (Nervous system disorders) | 4
Taste alteration (dysgeusia) (Nervous system disorders) | 8
Insomnia (Psychiatric disorders) | 6
Mood alteration - anxiety (Psychiatric disorders) | 7
Urinary frequency/urgency (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 23
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 30
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 3
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 4
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 5
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No